CLINICAL TRIAL: NCT03205774
Title: Effect of Positioning on Ultrasound Examination of the Gastric Antrum
Brief Title: Positioning and Ultrasound Examination of the Gastric Antrum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital Edouard Herriot (Other)
Responsible Party: Principal Investigator, Lionel Bouvet, MD, PhD, Hôpital Edouard Herriot
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: L16-190
Record Dates: First submitted 2017-06-28; First posted 2017-07-02 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Gastric Ultrasound

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Supine position (Sham Comparator): patient in supine position, lying on the back, turned in the right lateral decubitus and turned in the left lateral decubitus in a randomized way, after prolonged fasting and 10 min after free oral intake of water
  Interventions: Behavioral: 6 hours fasting and free oral intake of water
- 30° semirecumbent position (Sham Comparator): patient in semirecumbent position (head of the bed elevated to 30°), lying on the back, turned in the right lateral decubitus and turned in the left lateral decubitus in a randomized way, after prolonged fasting and 10 min after free oral intake of water
  Interventions: Behavioral: 6 hours fasting and free oral intake of water
- 45° semirecumbent position (Sham Comparator): patient in semirecumbent position (head of the bed elevated to 45°), lying on the back, turned in the right lateral decubitus and turned in the left lateral decubitus in a randomized way, after prolonged fasting and 10 min after free oral intake of water
  Interventions: Behavioral: 6 hours fasting and free oral intake of water
- 90° semirecumbent position (Sham Comparator): patient in semirecumbent position (head of the bed elevated to 90°), lying on the back, after prolonged fasting and 10 min after free oral intake of water
  Interventions: Behavioral: 6 hours fasting and free oral intake of water

INTERVENTIONS:
Behavioral: 6 hours fasting and free oral intake of water — Ultrasound examination of the gastric antrum are performed in volunteers after prolonged fasting and 10 min after oral intake of water. Volunteer should be lying on his/her back, right lateral decubitus position and left lateral decubitus position with randomization of the order.

SUMMARY:
The aim of this prospective study was to assess the effect of patient positioning on the ultrasound assessment of gastric contents.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 and 2 volunteers

Exclusion Criteria:

* Diabetes mellitus
* previous gastrointestinal surgery
* Medication affecting gastric motility
* digestive diseases, gastroparesis
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2018-01-20 (Actual); Study Completion 2018-01-20 (Actual)

PRIMARY OUTCOMES:
Change in ultrasound measurement of the antral cross sectional area according to the position | through study completion, an average of 20 min
  Ultrasound measurement of antral cross-sectional area
Change in qualitative ultrasound assessment of gastric contents according to the position | through study completion, an average of 20 min
  qualitative ultrasound assessment of gastric contents

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Femme Mère Enfant, Lyon, France